CLINICAL TRIAL: NCT02022995
Title: Investigation of Methylation of EGFR in the Response of the Cetuximab in Metastatic Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310053RIND
Record Dates: First submitted 2013-12-22; First posted 2013-12-30 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer Adenocarcinoma
Keywords: EGFR; cetuximab; colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with cetuximab treatment: Patients with cetuximab treatment
- Patients without cetuximab treatment: Patients without cetuximab treatment

SUMMARY:
Protein arginine methylation is an important process, which regulates diverse cellular functions including cell proliferation, RNA stability, DNA repair and gene transcription. Based on literature search, protein arginine methyltransferase (PRMT) indeed plays important roles in colon cancer pathophysiology. The PRMT expression level is involved in colon cancer patient's survival and has been suggested to be a prognostic marker in colon cancer patients. Recently, our group found a novel methylation on epidermal growth factor receptor (EGFR), which affected EGFR downstream signaling. investigators further observed the methylation event on EGFR not only regulated tumor growth in mouse xenograft model but also influenced cetuximab response in colon cancer cell lines. To further study the clinical correlation between EGFR methylation and cetuximab response, we propose to detect EGFR methylation level in paraffin embedded tissue samples from colorectal cancer patients with or without cetuximab treatment by IHC staining and analyze its correlation with cetuximab response. This study will provide an insight to the strategy of colorectal cancer therapy.

DETAILED DESCRIPTION:
Colorectal cancer is the third cause of cancer in the world. The recommended treatment of early stage (stage I and stage II) colorectal cancer is surgical removal, while the management of late stage (stage III and stage IV) colorectal cancer relies heavily on chemotherapy. Optimization of dosing and scheduling of chemotherapy agents are developed to improve response and survival rate of patients. Meanwhile, the rational targeting of molecular signaling pathways that are involved in the etiology of malignancies is currently one of the most promising strategies in novel anticancer drug development. Since first discovery of EGFR in 1962, EGFR family and its downstream signaling has become one of the most well characterized receptor tyrosine kinase system. In addition to their function in normal development, aberrant expression of EGFR is involved in abnormal cell proliferation, reduced apoptosis, cell migration, metastasis, angiogenesis and resistance to radiation and chemotherapy in cancer patients. Owing to the important role that EGFR plays in tumorigenesis, new classes of drugs that target EGFR, such as cetuximab, are among the most clinically advanced molecular-targeted therapies. The combination of EGFR monoclonal antibody with chemotherapy has shown efficacy in colorectal cancer treatment. However, the resistance of EGFR target therapy was recently observed due to complicated and different drug resistance mechanisms. Take EGFR monoclonal antibody, cetuximab, as an example, the response rate of cetuximab-plus-irinotecan therapy was about 23%. Some studies showed the resistance of EGFR to cetuximab is related to constitutive activation of mutant KRAS. However, more and more studies showed not all wild type KRAS patients response to cetuximab, while not all mutant Kras patients are refractory to cetuximab. These observations make it urgent to investigate the potential EGFR regulation mechanisms that may influence and predict the cetuximab response.

Epigenetic modifications, such as alterations in DNA methylation patterns and histone changes, play critical roles in human disease. Since identification of protein arginine methyltransferases (PRMTs), arginine methylation has been largely recognized and is under robust investigation. During arginine methylation process, PRMTs transfer methyl groups from S-adenosylmethionine (SAM) to guanidine nitrogenes of specific arginine residues on their target proteins. After arginine methylation, protein structure, protein-protein interaction, protein localization and enzyme activity are changed. As a result, diverse cellular functions including signal transduction, RNA processing, DNA repair and gene transcription are under regulation of arginine methylation. Recently, emerging evidences have shown links between dysfunction of arginine methylation and cancers. In prostate cancer, H4R3 methylation by PRMT predicts the risk of cancer recurrence; in Mixed Lineage Leukaemia (MLL), PRMT mediates transcriptional upregulation during cancer progression. Moreover, aberrantly high expression of PRMT is observed in tumor tissues of both breast and colorectal cancer and, notably, is associated with poor clinical outcomes in colorectal cancer patients. Given the importance of PRMT and EGFR in colorectal cancer development and progression, investigators tried to further investigate the relation between EGFR and PRMT in colorectal cancer pathophysiology.

In our preliminary data, investigators found PRMT can methylate EGFR, leading to up-regulation of EGFR signaling. The up-regulated EGFR signaling further triggered higher cell proliferation rate. In addition, cells with higher EGFR methylation level showed higher tumor growth ability in mice colorectal cancer xenograft model. Importantly, the cells with higher EGFR methylation level demonstrated higher cell growth rate in the presence of cetuximab in in vitro cell proliferation assay, suggesting that EGFR methylation may lead to resistance to cetuximab. In order to study the clinical correlation between EGFR methylation and cetuximab resistance, investigators propose to collect paraffin embedded tissue samples from patients with or without cetuximab treatment and analyze their EGFR methylation level. Investigators expect that patients with lower EGFR methylation level have higher improvement when treated with cetuximab compared to those without cetuximab treatment. In contrast, patients with higher EGFR methylation level showed poorer improvement when treated with cetuximab in comparison with patients without cetuximab treatment. By detecting EGFR methylation levels in these tissue samples and analyzing the correlation between EGFR methylation level and cetuximab response, investigators will provide an insight for prediction of cetuximab response in colorectal cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer stage IV

Exclusion Criteria:

* Age under 20 years old and over 80 years old Patient didn't have surgery in NTUH

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age between 20-80 years old Patient had surgery in NTUH
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
evaluate the overall survival of patients with PRMT (arginine methyltransferase) | 24 months

SECONDARY OUTCOMES:
evaluate the disease-free survival of patients with PRMT (arginine methyltransferase) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Been-Ren Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan